CLINICAL TRIAL: NCT04863482
Title: Safety of Laparoscopic ChOlecystectomy Performed by Trainee Surgeons With Different CHolangiographic Techniques
Acronym: SCOTCH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Università Politecnica delle Marche (Other)
Responsible Party: Principal Investigator, Monica Ortenzi, principal investigator, Università Politecnica delle Marche
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UPolitecnicaDM
Record Dates: First submitted 2021-04-12; First posted 2021-04-28 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-10

CONDITIONS: Cholecystitis; Gallstone
MeSH Terms: conditions — Cholecystitis; Gallstones

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Critical view of Safety (CVS-WL) (Active Comparator): Group CVS-WL (control group): the visualization of the biliary tree is achieved in white light, without the utilization of an intraoperative imaging technique, the CVS in white light was selected as the control group since it constitutes the actual recognized standard in clinical practice.
  Interventions: Procedure: IOC
- Intra-operative Cholangiography (IOC) (Experimental): Group IOC: the visualization of the biliary tree is achieved with the help of intraoperative cholangiography
  Interventions: Procedure: IOC
- Near-Infra Red Cholangiography (NIR-C) (Experimental): Group NIR-C: the visualization of the biliary tree is achieved with the help of near-infrared fluorescence cholangiography
  Interventions: Procedure: IOC

INTERVENTIONS:
Procedure: IOC — intra-operative cholangiography near-infrared fluorescence cholangiography
  Other Names: NIR-C

SUMMARY:
Laparoscopic cholecystectomy (LC) gained popularity among general surgeons in 1990s and rapidly become one of the most commonly performed procedures in digestive surgery, with more than one million cholecystectomies being performed in the United States per year. LC remains also one of the most commonly performed procedure by general surgeons during the training period. Even if previous report LC cases performed by surgical trainees (ST) are not associated with higher operative morbidity, the length of operative time is significantly increased when compared with that of LC cases performed by attending surgeons, due, most of all, to difficulties in identifying the anatomical structure, and this sometimes leads to an attending surgeon taking away the case from the trainee. Furthermore, despite the fact that LC has proven to be a safe procedure, the rate of common bile duct (BDI) injury still remains unacceptably high even in the hands of minimally invasive trained surgeons ranging from 0.2 to 1.5% in individual reports, much higher than initial reports, associated with significant morbidity and mortality, lower quality of life and increased costs, related to additional health care measures, loss of work days, and insurance claims. The aim of this study is to address which of the techniques now available could be addressed as the best option in a training setting to enhance the learning curve, to ideally build a safe cholecystectomy training program and virtually eliminate the risk of BDI due to anatomic misinterpretation during the training period.

DETAILED DESCRIPTION:
Study design The study will be a multicentre prospective observational study. Members of the Italian Society of Endoscopic Surgery [SICE] will be invited to participate. All participating centers will be required to register the study according to local regulations. Evidence of successful registration should be sent to your national network committee prior to beginning of data collection.

Rationale for Study Design Since to date there is no consensus on which is the best technique to correctly identify the anatomy of the Calot's triangle during LC performed by ST, this trial would aim to propose a standard technique to be used in this peculiar setting.

Potential Benefit for Patients In teaching hospitals and, more generally in a training setting, overcoming the problem of providing high surgical quality while educating ST can be challenging. This may change in the future if residents are able to better identify the anatomy with Intra-operative fluorescent cholangiography (IOIFC), shortening the learning curve and improving the safety profile of LC, that, in a clinical point of view, would translate into a shorter operative times and reduction of the potential risk of BDI.

Patient Risk There are no additional risks on the participation of this study as no additional procedures are being performed to clinical guidance. In accordance with standard care, patients shall receive written information regarding the index procedure.

Evaluated parameters i) Age ii) Sex iii) ASA scores iv) Preoperative work up v) Type of procedure (CVS-WL, NIFC, IOC) vi) Operative parameters (operative time, intraoperative complications) vii) BDI (according to the ATOM classification) viii) How the BDI was diagnosed intraoperatively ix) Duration of cholangiography x) Time needed to obtain a CVS xi) Post-operative outcomes (post-operative complications, late complications, need of readmission, length of hospital stay) xii) Surgeons' ease at performing the procedure (questionnaire on identification of anatomical structures, NASA task load test) xiii) Surgeons' satisfaction (visual analog scale)

Selection of Subjects Consecutive eligible patients will be recruited at the outpatient clinic in the participating center by the involved physician (surgeon). All patients fulfilling the above-mentioned criteria will be informed about the study by the physician. After consent is given, central data acquisition will take place web-based and patients will treated according to the study protocol.

Consent Potential participants will be counselled by a member of the research team directly involved with the study and who hold good clinical practice certification. Patients will be provided with written information and the consent form at the time of counselling with an opportunity to ask any questions. All patients participating in the study must hold capacity- this is an inclusion criteria and the absence of it an exclusion criteria.

Study procedures Critical view of Safety(CVS) The CVS has 3 requirements. First, the triangle of Calot must be cleared of fat and fibrous tissue. It does not require that the common bile duct be exposed. The second requirement is that the lowest part of the gallbladder be separated from the cystic plate, the flat fibrous surface to which the non peritonealized side of the gallbladder is attached. The cystic plate, which is sometimes referred to as the liver bed of the gallbladder, is part of the plate/sheath system of the liver. The third requirement is that 2 structures, and only 2, should be seen entering the gallbladder. Once these 3 criteria have been fulfilled, CVS has been attained). The rationale of CVS is based on a 2-step method for ductal identification that was and continues to be used in open cholecystectomy. First, by dissection in the triangle of Calot, the cystic duct and artery are putatively identified and looped with ligatures. Next, the gallbladder is completely dissected off the cystic plate, demonstrating that the 2 structures are the only structures still attached to the gallbladder. Time consumption and includes the period from the initial dissection and the obtaining of an acceptable view according to the previously described criteria in order to safely transect the cystic duct.

Intraoperative cholangiography (IOC)

IOC is performed after dissection of the cystic duct in a standardised manner, by cannulation of the cystic duct with a catheter using either a Kumar or Olsen grasper. Leakage is controlled by injecting saline prior to injection of iodine contrast means, according to the centre usual habits. A mobile X-ray C-arm system is used, and the monochrome X-ray image is shown on a separate screen. After satisfactory identification of the extra-hepatic biliary ducts, the intraoperative cholangiography is discontinued and the gallbladder is removed in a standardised manner. Time consumption includes the period from application of the Kumar/Olsen grasper until it is removed again after obtaining a satisfactory cholangiogram and the cystic duct is transected.

Near infrared cholangiography (NIR-C)

NIFC is performed injecting intravenously, 2.5-7.5 mg of indocyanine green (0.2 mg/kg) at the admission of the patients into the hospital, in patients admitted he same day of surgery, and at least 45 mins before the acquisition of the images. Indocyanine green rapidly binds to plasma proteins and is exclusively and entirely excreted by the hepatic parenchymal cells into the bile, starting within a few minutes after injection. During dissection, the fluorescence imaging mode is used when needed until critical view of safety is obtained. Before division of any tubular structure, the fluorescence imaging mode is routinely used again, and fluorescent angiography is performed by re-injecting the same dose of indocyanine green as initially used. After division of the cystic duct and artery, the fluorescence imaging mode is applied again to check for bile leakage. Time consumption and includes the period from the initial dissection and the obtaining of an acceptable CVS and transect the cystic duct.

Statistical analysis Descriptive statistics will be provided for all discrete variables in the form of rates and proportions with 95% confidence intervals. Continuous variables will be described by mean, standard deviation, median and range. Overall survival, disease free survival, local recurrence rate and metastasis rate will be estimated using the method of Kaplan Meier. Exploratory comparisons of discrete variables will be performed using a Chi-squared test, using continuity correction or Fisher's exact test. Continuous variables will be compared using a Student's t-test, or a non-parametric equivalent (Wilcoxon). All tests will be two sided with a p-value of less than 0.05 considered to indicate statistical significance. Data will be analysed according to intention-to treat principles.

Sample size Sample size was estimated using simulations for a superiority design. Assuming a success rate of 80% for the conventional intraoperative cholangiography, 90 % for the intraoperative fluorescent cholangiography and . This was done for a range of sample sizes. We then analysed each dataset to test whether intraoperative fluorescent cholangiography was no more than 10% inferior to conventional intraoperative cholangiography in a one-sided test applying a 5% level of significance. In conclusion, 60 patients in each group would yield a power of 90%.

Prior to data collection, assuming a baseline structure detection rate of 20%, 300 subjects per group was the estimated sample size needed to detect a 10% absolute increase (from 20 to 30%) in extrahepatic biliary structure visualization rates, with 95% confidence and 80% power. In addition to comparing structure detection rates between the 2 study arms, exploratory analysis was performed to identify potential effect modifiers like age, sex, body mass index (BMI), liver

Based on power calculations to demonstrate superiority of NBI over WLE for the endoscopic diagnosis of coeliac disease, 328 patients would be required in total (44 in each group): calculated using a significance level (alpha) 5%, power 1 (beta) 95%, %success in control (WLE) group 60% [25] and % success in experimental group (NBI) 91%.

The sample size has been considered with reference to (1) recruitment (2) adequately powered calculations to be conducted to address the outcomes including inter-observer variation.

Expected Duration of Trial The trial is expected to run for 6 months (time from first patient recruitment to last patient evaluation). Data analysis will take a maximum of 3 months after this time.

11. Ethics & Regulatory Approvals The trial will be conducted in compliance with the principles of the Declaration of Helsinki (1996), the principles of GCP and in accordance with all applicable regulatory requirements including but not limited to the Research Governance Framework and the Medicines for Human Use (Clinical Trial) Regulations 2004, as amended in 2006 and any subsequent amendments.

This study protocol will be submitted for local REC review in addition with patient information leaflet and consent form. The protocol/ any amendments will follow the local REC process. The chief investigator shall provide annual REC reports as required and will notify the REC at the end of the study.

If the study is ended prematurely, the Chief Investigator will notify the REC, including the reasons for the premature termination.

Data Handling

The Chief Investigator will act as custodian for the trial data. The following guidelines will be strictly adhered to:

All study data will be:

* Stored in line with the Medicines for Human Use (Clinical Trials) Amended Regulations 2006 and the Data Protection Act.
* archived in line with the Medicines for Human Use (Clinical Trials) Amended Regulations 2006 as defined in the Joint Clinical Trials Office Archiving SOP

ELIGIBILITY:
Inclusion Criteria:

* Patient scheduled for elective laparoscopic cholecystectomy
* Patient age ≥ 18 years
* Patient able to give consent to the procedure

Exclusion Criteria:

* Open cholecystectomy
* Emergency laparoscopic cholecystectomy
* Allergy towards iodine or indocyanine green
* Liver or renal insufficiency
* Thyrotoxicosis
* Pregnancy or lactation
* Legally incompetent for any reason
* Withdrawal of inclusion consent at any time
* Age outside inclusion range

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Time to obtain the CVS during laparoscopic cholecystectomy | operative period
  The primary objective is to compare NIFC, IOC and CVS-WL for identification of the junction between the cystic duct, the common hepatic duct and the CBD during LC performed by general surgery trainee always supported by an expert surgeon. The technique will be considered successful when the CVS will be achieved. The time to achieve the CVS will be recorded by an independent surgeon who will be present in the operative room during the procedure

SECONDARY OUTCOMES:
length of hospital stay | through study completion, an average of 1 year
  measured in days from the intervention to discharge
short term complications (reported with a descriptive name of scale and entered in an excel sheet) | up to 30 days from operation
  every unexpected event that will occur in the early post-operative period will be reported namely, the most likely that are thought to occur are bile leak, fever, pain
Operative time | operative period
  time from the first incision to trocars extraction
Intraoperative complications will be recorded namely as a descriptive variable and at the end of the study the frequency of each complication will be reported | operative period
  every unexpected event that will occur in the intra-operative period will be reported namely and at the end of the study frequencies of them will be provided
Need for conversion will be reported as a binomial variable and participants will be asked to feel the appropriate spaces with a 1 for yes and 0 for no, at the end the frequency of conversion occurrence will be provided | operative period
  Binomial scale
Causes for conversion will be reported as a descriptive variable and at the end of the study frequencies will be reported | operative period
  every event that will make conversion to open surgery necessary will be reported namely and at the end of the study frequencies of each of them will be provided
Type of BDI | operative period
  the type of IBD will be enlisted as nominal variables, the singular type of complication will be reported as frequencies
rate of BDI | operative period
  the occurrence of BDI will be reported and showed as a rate at the end of the study
Type of post-operative admission | immediate post-operative period
  recorded as a nominal variable and aimed to assess the necessity of an intensive care unit admission
Intensive care unit stay | up to 24 weeks
  measured as days spent in ICU unity

OTHER OUTCOMES:
Surgeon's satisfaction | operative period
  Surgeon's satisfaction will be measured with a visual analog scale (minimun value 0,maximum value 5) thet the operating surgeon will have to complete at the end of the operationeons' satisfaction will be assessed with a VAS analog scale that the operating
Surgeon's task load | operative period
  Surgeons will be asked to complete the NASA-TLX workload assessment questionnaire at the end of the operation

CONTACTS AND LOCATIONS:
Overall Officials: Monica Ortenzi, MD, Principal Investigator — Università Politecnica delle Marche
Locations (1):
- Università Politecnica delle Marche, Clinica Chirurgica, Ancona, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Way LW, Stewart L, Gantert W, Liu K, Lee CM, Whang K, Hunter JG. Causes and prevention of laparoscopic bile duct injuries: analysis of 252 cases from a human factors and cognitive psychology perspective. Ann Surg. 2003 Apr;237(4):460-9. doi: 10.1097/01.SLA.0000060680.92690.E9. PMID 12677139
- [Background] Pucher PH, Brunt LM, Fanelli RD, Asbun HJ, Aggarwal R. SAGES expert Delphi consensus: critical factors for safe surgical practice in laparoscopic cholecystectomy. Surg Endosc. 2015 Nov;29(11):3074-85. doi: 10.1007/s00464-015-4079-z. Epub 2015 Feb 11. PMID 25669635
- [Background] CHERRICK GR, STEIN SW, LEEVY CM, DAVIDSON CS. Indocyanine green: observations on its physical properties, plasma decay, and hepatic extraction. J Clin Invest. 1960 Apr;39(4):592-600. doi: 10.1172/JCI104072. No abstract available. PMID 13809697
- [Background] Blom EM, Verdaasdonk EG, Stassen LP, Stassen HG, Wieringa PA, Dankelman J. Analysis of verbal communication during teaching in the operating room and the potentials for surgical training. Surg Endosc. 2007 Sep;21(9):1560-6. doi: 10.1007/s00464-006-9161-0. Epub 2007 Feb 7. PMID 17285367
- [Background] Strasberg SM, Hertl M, Soper NJ. An analysis of the problem of biliary injury during laparoscopic cholecystectomy. J Am Coll Surg. 1995 Jan;180(1):101-25. No abstract available. PMID 8000648
- [Background] Ishizawa T, Bandai Y, Kokudo N. Fluorescent cholangiography using indocyanine green for laparoscopic cholecystectomy: an initial experience. Arch Surg. 2009 Apr;144(4):381-2. doi: 10.1001/archsurg.2009.9. No abstract available. PMID 19380655
- [Background] Photi ES, El-Hadi A, Brown S, Swafe L, Ashford-Wilson S, Barwell J, Koopmans I, Lewis MPN. The Routine Use of Cholangiography for Laparoscopic Cholecystectomy in the Modern Era. JSLS. 2017 Jul-Sep;21(3):e2017.00032. doi: 10.4293/JSLS.2017.00032. PMID 28951654
- [Background] Ludwig K, Bernhardt J, Steffen H, Lorenz D. Contribution of intraoperative cholangiography to incidence and outcome of common bile duct injuries during laparoscopic cholecystectomy. Surg Endosc. 2002 Jul;16(7):1098-104. doi: 10.1007/s00464-001-9183-6. Epub 2002 Apr 9. PMID 12165830
- [Background] Flum DR, Koepsell T, Heagerty P, Sinanan M, Dellinger EP. Common bile duct injury during laparoscopic cholecystectomy and the use of intraoperative cholangiography: adverse outcome or preventable error? Arch Surg. 2001 Nov;136(11):1287-92. doi: 10.1001/archsurg.136.11.1287. PMID 11695975
- [Background] Polat FR, Abci I, Coskun I, Uranues S. The importance of intraoperative cholangiography during laparoscopic cholecystectomy. JSLS. 2000 Apr-Jun;4(2):103-7. PMID 10917115
- [Background] Lill S, Rantala A, Pekkala E, Sarparanta H, Huhtinen H, Rautava P, Gronroos JM. Elective laparoscopic cholecystectomy without routine intraoperative cholangiography: a retrospective analysis of 1101 consecutive cases. Scand J Surg. 2010;99(4):197-200. doi: 10.1177/145749691009900403. PMID 21159587
- [Background] Ding GQ, Cai W, Qin MF. Is intraoperative cholangiography necessary during laparoscopic cholecystectomy for cholelithiasis? World J Gastroenterol. 2015 Feb 21;21(7):2147-51. doi: 10.3748/wjg.v21.i7.2147. PMID 25717250
- [Background] Takada T, Strasberg SM, Solomkin JS, Pitt HA, Gomi H, Yoshida M, Mayumi T, Miura F, Gouma DJ, Garden OJ, Buchler MW, Kiriyama S, Yokoe M, Kimura Y, Tsuyuguchi T, Itoi T, Gabata T, Higuchi R, Okamoto K, Hata J, Murata A, Kusachi S, Windsor JA, Supe AN, Lee S, Chen XP, Yamashita Y, Hirata K, Inui K, Sumiyama Y; Tokyo Guidelines Revision Committee. TG13: Updated Tokyo Guidelines for the management of acute cholangitis and cholecystitis. J Hepatobiliary Pancreat Sci. 2013 Jan;20(1):1-7. doi: 10.1007/s00534-012-0566-y. PMID 23307006
- [Background] Sajid MS, Leaver C, Haider Z, Worthington T, Karanjia N, Singh KK. Routine on-table cholangiography during cholecystectomy: a systematic review. Ann R Coll Surg Engl. 2012 Sep;94(6):375-80. doi: 10.1308/003588412X13373405385331. PMID 22943325
- [Background] Soper NJ, Dunnegan DL. Routine versus selective intra-operative cholangiography during laparoscopic cholecystectomy. World J Surg. 1992 Nov-Dec;16(6):1133-40. doi: 10.1007/BF02067079. PMID 1455885
- [Background] Pesce A, Latteri S, Barchitta M, Portale TR, Di Stefano B, Agodi A, Russello D, Puleo S, La Greca G. Near-infrared fluorescent cholangiography - real-time visualization of the biliary tree during elective laparoscopic cholecystectomy. HPB (Oxford). 2018 Jun;20(6):538-545. doi: 10.1016/j.hpb.2017.11.013. Epub 2017 Dec 29. PMID 29292071
- [Background] Pesce A, Piccolo G, La Greca G, Puleo S. Utility of fluorescent cholangiography during laparoscopic cholecystectomy: A systematic review. World J Gastroenterol. 2015 Jul 7;21(25):7877-83. doi: 10.3748/wjg.v21.i25.7877. PMID 26167088
- [Background] Agnus V, Pesce A, Boni L, Van Den Bos J, Morales-Conde S, Paganini AM, Quaresima S, Balla A, La Greca G, Plaudis H, Moretto G, Castagnola M, Santi C, Casali L, Tartamella L, Saadi A, Picchetto A, Arezzo A, Marescaux J, Diana M. Fluorescence-based cholangiography: preliminary results from the IHU-IRCAD-EAES EURO-FIGS registry. Surg Endosc. 2020 Sep;34(9):3888-3896. doi: 10.1007/s00464-019-07157-3. Epub 2019 Oct 7. PMID 31591654
- [Background] Liu Y, Peng Y, Su S, Fang C, Qin S, Wang X, Xia X, Li B, He P. A meta-analysis of indocyanine green fluorescence image-guided laparoscopic cholecystectomy for benign gallbladder disease. Photodiagnosis Photodyn Ther. 2020 Dec;32:101948. doi: 10.1016/j.pdpdt.2020.101948. Epub 2020 Aug 6. PMID 32771612
- [Background] Quaresima S, Balla A, Palmieri L, Seitaj A, Fingerhut A, Ursi P, Paganini AM. Routine near infra-red indocyanine green fluorescent cholangiography versus intraoperative cholangiography during laparoscopic cholecystectomy: a case-matched comparison. Surg Endosc. 2020 May;34(5):1959-1967. doi: 10.1007/s00464-019-06970-0. Epub 2019 Jul 15. PMID 31309307
- [Background] Lehrskov LL, Westen M, Larsen SS, Jensen AB, Kristensen BB, Bisgaard T. Fluorescence or X-ray cholangiography in elective laparoscopic cholecystectomy: a randomized clinical trial. Br J Surg. 2020 May;107(6):655-661. doi: 10.1002/bjs.11510. Epub 2020 Feb 14. PMID 32057103
- [Background] Sariego J, Spitzer L, Matsumoto T. The "learning curve" in the performance of laparoscopic cholecystectomy. Int Surg. 1993 Jan-Mar;78(1):1-3. PMID 8473074
- [Background] Hawasli A, Lloyd LR. Laparoscopic cholecystectomy. The learning curve: report of 50 patients. Am Surg. 1991 Aug;57(8):542-4; discussion 545. PMID 1834000
- [Background] Moore MJ, Bennett CL. The learning curve for laparoscopic cholecystectomy. The Southern Surgeons Club. Am J Surg. 1995 Jul;170(1):55-9. doi: 10.1016/s0002-9610(99)80252-9. PMID 7793496
- [Background] Cagir B, Rangraj M, Maffuci L, Herz BL. The learning curve for laparoscopic cholecystectomy. J Laparoendosc Surg. 1994 Dec;4(6):419-27. doi: 10.1089/lps.1994.4.419. PMID 7881146
- [Background] Fingerhut A, Dziri C, Garden OJ, Gouma D, Millat B, Neugebauer E, Paganini A, Targarona E. ATOM, the all-inclusive, nominal EAES classification of bile duct injuries during cholecystectomy. Surg Endosc. 2013 Dec;27(12):4608-19. doi: 10.1007/s00464-013-3081-6. Epub 2013 Jul 27. PMID 23892759